CLINICAL TRIAL: NCT02551705
Title: Functional Imaging of Social Cognition in Premanifest Huntington's Disease
Acronym: FISCIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Jan Van den Stock, Post-doctoral researcher, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S58457
Record Dates: First submitted 2015-09-07; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Functional Neuroimaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- functional Imaging mutation carrier (Experimental): Premanifest mutation carrier, behavioral and neural emotional memory processing
  Interventions: Other: functional Imaging
- functional Imaging non-carrier (Active Comparator): non-carrier family member, behavioral and neural emotional memory processing
  Interventions: Other: functional Imaging

INTERVENTIONS:
Other: functional Imaging — Brain responses associated with emotional memory will be investigated

SUMMARY:
Huntington's disease (HD) is a genetic progressive fatal neurodegenerative disorder. In the western world it affects 5-10 persons per 100000. The main brain changes include the loss of brain cells in subcortical structures. The symptoms of HD include involuntary movements, cognitive deterioration and behavioural disturbances. It has been shown that changes in emotion comprehension occur before the onset of the motor symptoms (preHD). This deficit in perception of emotions has been primarily investigated by means of facial expressions. However, emotions can also be expressed through body language. Here, the investigators propose to investigate whether the emotion comprehension deficit in preHD also includes body language comprehension.

DETAILED DESCRIPTION:
The investigators will perform a detailed evaluation of body language comprehension abilities in persons that carry the genetic mutation causing HD, but who do not show any movement symptoms yet. In addition, the associated changes in brain structure and function will be studied. The aim is to perform the study with the same group of participants who participated in a recent study carried on by this research group, in which the functional brain changes associated with increased irritability were investigated. This will allow to relate emotion experience with emotion perception. The results of the study may provide a target to further develop therapeutic interventions and aid caregivers of preHD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Huntington's disease positive genotype and non-carrier siblings

Exclusion Criteria:

* visible chorea
* MRI contra-indications
* major neurological/psychiatric comorbidity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Significant group differences in brain activation for perceiving emotional vs neutral faces by following random effects analyses | 6 months
  Significant group differences in beta-values for the contrast emotional faces vs neutral faces following general linear model parameter estimates